CLINICAL TRIAL: NCT04876118
Title: Feasibility Study of CoolSculpting Effects on Cellulite Appearance
Brief Title: Effects on Cellulite Appearance
Acronym: EFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA20-002
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fat Reduction (Experimental): The treatments are designed to see if the appearance of cellulite can be reduced on the outer thigh.
  Interventions: Device: The ZELTIQ System

INTERVENTIONS:
Device: The ZELTIQ System — The CoolSculpting machine will be used to perform the treatments.

SUMMARY:
Evaluate the safety and feasibility effecting the appearance of cellulite on the thigh using CoolSculpting.

ELIGIBILITY:
Inclusion Criteria

* Female subjects > 22 years of age and < 65 years of age.
* Subject has clearly visible cellulite on the intended treatment area (thighs), which in the Investigator's opinion, may benefit from the treatment.
* Subject has not had weight change exceeding 5% in the preceding month.
* Subject agrees to maintain her weight (i.e., within 5%) by not making any major changes in diet or exercise routine during the course of the study.
* Subject has read and signed a written informed consent form.

Exclusion Criteria

* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction, body contouring, cellulite reduction and/or skin tightening procedure in the area of intended treatment within the past 4 months.
* Presence of significant suntan in the thighs.
* Inability to avoid sun exposure in the thighs.
* Subject has a history of hernia in or adjacent to the areas to be treated.
* Subject needs to administer or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, cold agglutinin disease, or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the Investigator's opinion may increase the subject's risk of bruising.
* Subject has known sensitivity or allergy to isopropyl alcohol and propylene glycol.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites, that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, implants (e.g. buttock implants), or drug delivery system.
* Subject is pregnant or intending to become pregnant during the study period (in the next 9 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the Investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Zeltiq Aesthetics
Locations (6):
- United States (6):
  - Investigate MD, Scottsdale, Arizona
  - Rebecca Fitzgerald, MD Dermatology, Los Angeles, California
  - Sasaki Advanced Aesthetics Medical Center, Pasadena, California
  - Innovation Research Center, Pleasanton, California
  - Laser and Skin Surgery Center of Northern California, Sacramento, California
  - Aesthetic Solutions, P.A., Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CoolSculpting of the Thigh: Participants received up to 2 CoolSculpting treatments of the thigh performed at up to 6 weeks apart.
Period: Overall Study
Arm/Group | CoolSculpting of the Thigh
Started | 97
Received at Least 1 Study Treatment | 97
Per Protocol Population | 74
Completed | 82
Not Completed | 15
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 treatment.
Arm/Group | CoolSculpting of the Thigh
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 82
  Race: Black or African American | 3
  Race: Asian | 5
  Race: American Indian or Alaska Native | 1
  Race: Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Photographs Correctly Identified by Blinded Reviewers From the Independent Physician Reviewer Panel
Description: Photographs of the treatment area taken at baseline and 12-weeks after final treatment were assessed for visual changes. Reported here is the mean percentage (%) of correct baseline identification of images by the blinded independent reviewers.
Time Frame: Week 12 post final treatment (up to 24 weeks after first treatment)
Population: Per Protocol population consisted of all treated participants who 2 treatments, and weight change of no more than 5% of total body weight at the time the assessments were performed compared to the weight obtained at the first treatment visit. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Number; unit: % of images identified correctly
Arm/Group | CoolSculpting of the Thigh
Number analyzed (Participants) | 73
% of images identified correctly | 55.7

2. Secondary Outcome: Number of Participants With Device and/or Procedure Related Adverse Events (AEs) and Device-related Serious Adverse Events (SADEs)
Description: An AE was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, whether or not considered related to treatment. A serious AE was an AE that resulted in death, serious deterioration in health, permanent impairment of a body structure/function, was life-threatening, required hospitalization or medical/surgical intervention, led to fetal distress or death, congenital abnormality, or birth defect. An adverse devise effect (ADE) was any sign, symptom, or disease determined by the Investigator to have a causal relationship or possible causal relationship with the investigational device, including any AE resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the device or from use error or intentional misuse of the device. A SADE was an ADE that resulted in any of the consequences characteristic of a serious AE.
Time Frame: Baseline up to 36 weeks post final treatment (up to 42 weeks from first treatment)
Population: The Safety Population consisted of all enrolled participants who received at least 1 treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting of the Thigh
Number analyzed (Participants) | 97
Participants
  Device and/or Procedure Related AEs | 3
  SADEs | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 36 weeks post final treatment (up to 42 weeks from first treatment)
Description: The Safety Population consisted of all enrolled participants who received at least 1 treatment.
Arm/Group | CoolSculpting of the Thigh
All-Cause Mortality (participants affected / at risk) | 0/97
Serious Adverse Events (participants affected / at risk) | 4/97
Other Adverse Events (participants affected / at risk) | 11/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CoolSculpting of the Thigh (N=97)
Urinary Tract Infection (Renal and urinary disorders) | 1
Food Poisoning (Gastrointestinal disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Atypical lump of cells in left breast (Reproductive system and breast disorders) | 1
Fever (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CoolSculpting of the Thigh (N=97)
Reaction post COVID-19 booster (General disorders) | 1
Broken foot (Musculoskeletal and connective tissue disorders) | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1
Right arm fracture (Musculoskeletal and connective tissue disorders) | 1
COVID-19 (Infections and infestations) | 3
Herpes Zoster (Shingles) (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Contour irregularity (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT04876118/Prot_SAP_000.pdf